CLINICAL TRIAL: NCT01694732
Title: Efficacy of Varenicline Associated With Intensive Counselling Versus Placebo of Varenicline Associated With Intensive Counselling on Smoking Cessation at the Acute Phase of an Exacerbation of Chronic Obstructive Pulmonary Disease (COPD). A Multicenter Randomized Double-blind Trial
Brief Title: Efficacy of Varenicline on Smoking Cessation at the Acute Phase of an Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: SAVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAVE RB11-135; RB 11-135 (Registry Identifier: RB 11-135)
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD Exacerbation; Smoking
Keywords: Chronic obstructive pulmonary disease; Varenicline; Smoking cessation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline with counselling (Experimental): Active varenicline associated with intensive smoking cessation counselling
  Interventions: Drug: Varenicline
- Placebo with counselling (Placebo Comparator): Placebo of varenicline associated with intensive smoking cessation counselling
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Varenicline
  Arms: varenicline with counselling
Drug: placebo
  Arms: Placebo with counselling

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic inflammatory disease of the bronchi with an increasing prevalence. By 2020, the mortality related to COPD is expected to become the 3rd leading death worldwide. COPD is caused by smoking in approximately 90 % of the cases. Nevertheless, COPD remains under-diagnosed and more than half of patients remain active smokers. Brittany is the second region of France facing an abnormal high death rate related to COPD. Smoking cessation is the most effective therapeutic approach to reduce the evolution of the disease, the frequency of the exacerbations and the the mortality. Besides, smoking cessation is associated with a reduced risk of cardiovascular events and cancer. Given the COPD patients' strong addiction, smoking cessation is not easily obtained in such population. Furthermore, smoking cessation has been underestimated in several studies. Most of these studies evaluated various methods of smoking cessation in COPD patients performed after an exacerbation, which has a hospitalization related mortality of approximately 10%. Thus, there is an urgent need to find effective pharmacotherapies to help COPD patients to cease smoking. Varenicline, a partial agonist at a4ß2 nicotinic acetylcholine receptors is reported to be one of the most effective pharmacotherapies for smoking cessation. However, it has never been evaluated at the acute phase of an exacerbation of COPD requiring hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients smokers (= 10 cigarettes per day in the last year)
* Affected by a chronic obstructive pulmonary disease.
* Presenting a recent exacerbation having led to at least a 24-hour hospitalization in pneumology or intensive care unit.
* Inclusion during hospitalization.
* Motivated to quit smoking
* Able to understand the information and give a written consent.
* Available for a follow-up of 1 year.

Exclusion Criteria:

* Refusal or unable to consent.
* Unaffiliated or not entitled to the National Health Insurance Coverage.
* Absence of a chronic obstructive pulmonary disease according to the criteria ATS / ERS.
* presenting a contraindication to the pharmacotherapy (i.e. the active substance: tartrate of varénicline or one of the excipients)
* actively participating in other smoking cessation trials.
* Pregnancy: declared or planned in 14 months.
* breastfeeding.
* Women old enough to procreate without reliable contraception.
* History of anorexia nervosa or bulimia.
* History of a severe depression and having required a medicinal treatment in 5 years.
* History of 2 or several episodes of severe depression and having required a medicinal treatment.
* Personal or family History of suicide attempt.
* History or current presence of dementia, a bipolar disease, a psychosis, a panic attack.
* Taken by psychotropic medicines in the inclusion excepted those prescribed to hypnotic aim and antidepressant medicine of the class of the inhibitors of the recapture of the sérotonine prescribed for a not severe depression
* Presence of a depression detected by means of the questionnaire HAD (not inclusion if the total of the sub-scale D is > 8 or if the total of scales A + D is > 16) and/or PHQ-9 (not inclusion if score > 9).
* SGOT or SGPT > 2 fold upper limit of normal, the hepatic cirrhosis, the acute hepatitis.
* Renal insufficiency (clearance of the creatinine < 30 ml / min according to the formula of Cockcroft).
* Excessive consumption of alcohol (more than 21 glasses a week for the men, more than 14 glasses of wines a week to them Women).
* Use of marijuana or other forms of tobacco during the study.
* Use of other stimulant drugs (ephedrine, phenylephrine) or appetite suppressants during the study.
* Life expectancy of ≤ 12-months (ex: patients affected by a chronic disease in terminal phase).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To demonstrate an increase in smoking abstinence rate | 12 months
  To demonstrate that in smokers with COPD hospitalized for an exacerbation early initiation of a pharmacotherapy by varenicline during 12 weeks is associated with a higher rate of long-term smoking abstinence measured in 1 year compared to placebo.

SECONDARY OUTCOMES:
Estimate the tolerance of the varenicline | 3 months
  Evaluate the side effects of varenicline after 3 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Francis COUTURAUD, Pr, Principal Investigator — University hospital of Brest
Locations (13):
- France (13):
  - CHU Angers, Angers, France
  - Hôpital HIA Clermont Tonnerre, Brest, France
  - Cavale Blanche Hospital, Brest, France
  - Laennec Hospital, Nantes, France
  - Caremeau Hospital, Nîmes, France
  - Hotel Dieu Hospital, Paris, France
  - HEGP Hospital, Paris, France
  - Poitiers Hospital, Poitiers, France
  - Cornouaille Hospital, Quimper, France
  - Pontchaillou, Rennes, France
  - Saint Brieuc Hospital, Saint-Brieuc, France
  - Bretonneau Hospital, Tours, France
  - CHRU Lille, Lille

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Le Mao R, Tromeur C, Paleiron N, Sanchez O, Gagnadoux F, Jouneau S, Magnan A, Hayem-Vannimenus C, Dansou A, Proust A, Dion A, Larhantec G, Brestec AL, Dewitte JD, Roche N, Leroyer C, Couturaud F. Effect of Early Initiation of Varenicline on Smoking Cessation in COPD Patients Admitted for Exacerbation: The Save Randomized Clinical Trial. COPD. 2020 Feb;17(1):7-14. doi: 10.1080/15412555.2019.1703928. Epub 2019 Dec 19. PMID 31854207